CLINICAL TRIAL: NCT05050838
Title: Prone Positioning for Brain-injured Patients With Severe ARDS (ProBrain)
Acronym: ProBrain
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: CE_20181218_3_CG
Record Dates: First submitted 2021-09-09; First posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Cerebral Blood Flow
Keywords: Prone Position; Acute Respiratory Distress Syndrome; Intracranial Pressure
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Transcranial Doppler (TCD) — TCD ultrasonography is based on the principle of the Doppler effect. According to this principle, ultrasound waves emitted from the Doppler probe are transmitted through the skull and reflected by moving red blood cells within the intracerebral vessels. The difference in the frequency between the emitted and reflected waves, referred to as the "Doppler shift frequency," is directly proportional to the speed of the moving red blood cells (blood flow).
  Cerebral blood flow (in cm/s) of the middle cerebral artery will be measured with TCD in blood-injured ARDS patients before and one hour after prone positioning (normal ranges: 48 to 72 cm/s).

SUMMARY:
Prone position (PP) is a key component to treat hypoxemia in patients with severe acute respiratory distress syndrome (ARDS). However, most studies evaluating PP effects in patients with ARDS exclude those with brain-injuries without providing any medical evidence. This prospectice observational study aimed to investigate if prone positioning leads to significant modification of cerebral perfusion in brain-injured patients with ARDS.

ELIGIBILITY:
Inclusion Criteria:

* adult's patients suffering from brain injuries
* patients neurologically monitored with TCD
* patients requiring prone position for severe ARDS

Exclusion Criteria:

* pregnant women
* patients with contrindication to prone position

Ages: 18 Years to 95 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Brain-injured patients with ARDS requirering prone positioning
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Cerebral Blood Flow | 1 hour
  Cerebral Blood Flow measurement before and after prone positioning

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Fondation Adolphe de Rothschild, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No